CLINICAL TRIAL: NCT04042571
Title: Permanent Cerebral Oxymetry Monitoring for Early Diagnosis and Treatment of Delayed Vasospasm After Subarachnoid Hemorrhage
Acronym: COMOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/34
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Intracranial oxymetry; Subarachnoid Hemorrhage; Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral oxymetry monitoring (NIRS) (Experimental): Cerebral oxymetry (NIRS) -by rSO2 measurement - in order to detect vasospasm in patient with severe subarachnoid hemorrhage compare to standard monitoring tools
  Interventions: Device: Cerebral oxymetry monitoring (NIRS)

INTERVENTIONS:
Device: Cerebral oxymetry monitoring (NIRS) — Near-InfraRed Spectroscopy (NIRS) is a non-invasive method measuring tissue oxygenation by regional saturation of capillary-oxygenated hemoglobin (rSO2). Starting on day 4 after aneurismal rupture NIRS electrods will be placed and maintained until day 12 permanently and blindly recording rSO2. Patients will be monitored following daily practice recommandations inclunding vasospasm detection and treatment.

SUMMARY:
Transcranial Doppler ultrasound (TCD) monitoring and CT-scanner perfusion are useful but imperfect tools to identify vasospasm and allow intervention to avoid infarction.

Permanent monitoring of cerebral tissue oximetry (rSO2) by NIRS, a noninvasive method could allow better vasospasm detection.

This study will evaluate diagnostic accuracy of cerebral oxymetry (NIRS) -by rSO2 measurement - in order to detect vasospasm in patient with severe subarachnoid hemorrhage compare to standard monitoring tools.

DETAILED DESCRIPTION:
Delayed vasospasm is a serious complication of aneurismal subarachnoid haemorhage (SAH) significantly influencing morbidity and mortality. Mostly observed between days 4 and 10 after aneurismal rupture, its incidence is higher in cases of severe SAH. Vasospasm strongly affects prognisis generating delayed cerebral ischemia.

Clinical deterioration (focal neurological deficit) is the best way to detect severe vasospasm. Unfortunately, most of severe SAH are intubated and sedated prohibiting neurological evaluation. In these frequent situations, Transcranial Doppler (TCD), clinical and biological monitoring, CT-scanner (angio-CT and Perfusion-CT), MRI and cerebral angiography are routinely used to detect vasospasm. Yet, these tools have imperfect sensitivity and specificty delaying diagnosis and treatment.

Near-InfraRed Spectroscopy (NIRS) is a non-invasive method measuring tissue oxygenation by regional saturation of capillary-oxygenated hemoglobin (rSO2). This technology demonstrated ability to measure cerebral oxygenation and has previously been reported to monitor carotid and pediatric surgery. To date a few studies also reported NIRS monitoring feasability in post-SAH vasospasm. Our aim is here to evaluate NIRS monitoring for the diagnosis of vasospasm in severe SAH.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age ≥ 18 years
* HSA of aneurysmal etiology less than 4 days before inclusion diagnosed by clinical presentation and emergency imaging
* HSA "severe" defined according to the WFNS ≥ III
* Intubated-ventilated patient or any other reason preventing a contributing neurological examination
* Affiliate or beneficiary of a social security scheme
* Free, informed and written consent signed by the representative

Exclusion Criteria:

* Age <18 years
* Significant vasospasm as soon as the detection was detected on the initial imaging
* Possible Neurological Surveillance
* Patient in limitation of active therapeutics or with high probability of soon limitation of active therapeutics
* Intra-parenchymal frontal haematoma limiting the quality of measurement, diagnosed on imaging (Less than 25mm deep from the skin)
* Patient in limitation of active therapeutics or with high probability of soon limitation of active therapeutics
* Adhesive allergy to measuring patches
* Patient under guardianship or safeguard of justice
* Refusal of legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Permanent measurement of cerabral oxymetry (rSO2) by NIRS system | From day 4 to day 12 post aneurysmal subarachnoid hemorrhage
  Difference between NIRS basal measurement entre la mesure basale du NIRS (NIRS average on the first hour of recording respectively on the left and right) and the NIRS measurement during the follow-up (lowest mean NIRS observed over one hour in patients without vasospasm diagnosed by the reference test or mean NIRS observed over the hour.

SECONDARY OUTCOMES:
Severity of angiographic spasm | Day 8 post aneurysmal subarachnoid hemorrhage
  Not significant (<50%) Significant (>50%) Severe.
Pti02 value | Day 4 post aneurysmal subarachnoid hemorrhage
  Pti02 value (mm Hg)
Pti02 value | Day 8 post aneurysmal subarachnoid hemorrhage
  Pti02 value (mm Hg)
Pti02 value | Day 12 post aneurysmal subarachnoid hemorrhage
  Pti02 value (mm Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France